CLINICAL TRIAL: NCT05334797
Title: The Effect of Hot Application on Shoulder Pain and Analgesic Use After Laparoscopic Upper Abdominal Surgery
Brief Title: The Effect of Hot Application on Post Laparoscopic Shoulder Pain and Analgesic Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Derya Gezer, Assistant Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PLSP
Record Dates: First submitted 2022-04-09; First posted 2022-04-19 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Pain, Shoulder
Keywords: postlaparoscopic; shoulder pain; analgesic; Hot application
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hot application (Experimental): After the patients come to the service after the surgery, a thermophore filled with hot water will be placed on the patient's shoulder according to the presence of shoulder pain and it will be ensured that he stays for 15 minutes. Pain assessment will be done before and after the application. However, 0-2-4-8-12-24. Routine pain assessment will be done at In addition, the type, route, effect and amount of analgesic done in this process will also be recorded. Response evaluation will follow. Response evaluation will follow. Hot application will be applied to every shoulder pain reported by the patients.
  Interventions: Other: hot application
- control group (No Intervention): First, an individual information form will be filled in for the control group patients who meet the sampling criteria. 0-2-4-8-12-24 after the patients come to the service after the surgery. Routine pain assessment will be done at In addition, the type, route, effect and amount of analgesic done in this process will also be recorded. Response evaluation will follow.

INTERVENTIONS:
Other: hot application — a thermophore filled with hot water will be placed on the patient's shoulder according to the presence of shoulder pain and it will be ensured that he stays for 15 minutes.
  Arms: Hot application

SUMMARY:
The aim of this study; To evaluate the effect of hot application on postlaparoscopic shoulder pain and analgesic use in patients undergoing upper laparoscopic surgery in general surgery.

DETAILED DESCRIPTION:
Among the advantages of laparoscopic surgery; smaller incisions, less postoperative pain, less need for analgesia, shorter hospital stay, earlier return to normal activities and lower morbidity. However, laparoscopic surgery is associated with postoperative shoulder pain, which is rarely seen in open surgeries. The precise mechanism of postlaparoscopic shoulder pain (PLOA) is unclear, but it is believed that the carbon dioxide remaining after laparoscopic surgery causes shoulder pain by causing irritation of the phrenic nerve. In some cases, PLOA may cause more discomfort to the patient than incisional pain.

Hot application is an effective method used to relieve pain. Hot application activates the gate control mechanism, stimulating tactile receptors, reducing ischemic pain with vasodilation, removing metabolic wastes, increasing the release of endorphins, eliminating muscle spasm, reducing effects such as pressure, stretching and hypoxia on nerve endings as a result of changes in the viscoelastic properties of tissues, raising the pain threshold, It reduces or relieves pain by sedating and creating relief in the patient.

Hot application is easy to use, inexpensive, requires no prior application, and has minimal adverse side effects when used correctly. Heat sources include a hot water heater, an electric heating pad, a warm blanket, and a warm bath or shower. In addition to being used as a pain reliever, heat is used to relieve chills or shivering, reduce joint stiffness, reduce muscle spasm, and increase connective tissue extensibility.

In the study of Mohamed et al., in which they examined the effect of hot application and early mobilization on shoulder pain, in the experimental group patients who received hot application; Postoperative shoulder pain was found to be significantly less than the control group at different evaluation times at 4 hours after surgery and at 6, 12 and 24 hours (p<0.001).

ELIGIBILITY:
Inclusion Criteria:

1. Agreeing to participate in the research,
2. Having undergone laparoscopic abdominal surgery
3. Those who have no previous history of surgery

Exclusion Criteria:

1. Those who did not agree to participate in the research
2. Those who have had previous abdominal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
change of pain | 24 hours
  Numerical Pain Rating Scale (NRS) The form used by Williamson & Hoggart (2005) to assess pain, patients will be asked to select a number from 0 to 10 that best describes their current pain. 0 means no pain and 10 means severe pain. It will be scored as no pain (0), mild pain (1-3), moderate (4-7) and severe pain (8-10).
analgesic consumption | 24 hours
  analgesic consumption form

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus Universty, Mersin, Tarsus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Results about the effect of hot application on pain and analgesic use will be shared. however, personal information will not be shared.

REFERENCES:
- [Background] Grace PA, Quereshi A, Coleman J, Keane R, McEntee G, Broe P, Osborne H, Bouchier-Hayes D. Reduced postoperative hospitalization after laparoscopic cholecystectomy. Br J Surg. 1991 Feb;78(2):160-2. doi: 10.1002/bjs.1800780209. PMID 1826624
- [Background] Valla JS, Limonne B, Valla V, Montupet P, Daoud N, Grinda A, Chavrier Y. Laparoscopic appendectomy in children: report of 465 cases. Surg Laparosc Endosc. 1991 Sep;1(3):166-72. PMID 1669397
- [Background] Nieboer TE, Johnson N, Lethaby A, Tavender E, Curr E, Garry R, van Voorst S, Mol BW, Kluivers KB. Surgical approach to hysterectomy for benign gynaecological disease. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD003677. doi: 10.1002/14651858.CD003677.pub4. PMID 19588344
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Mouton WG, Bessell JR, Otten KT, Maddern GJ. Pain after laparoscopy. Surg Endosc. 1999 May;13(5):445-8. doi: 10.1007/s004649901011. PMID 10227938
- [Background] Fredman B, Jedeikin R, Olsfanger D, Flor P, Gruzman A. Residual pneumoperitoneum: a cause of postoperative pain after laparoscopic cholecystectomy. Anesth Analg. 1994 Jul;79(1):152-4. PMID 8010427
- [Background] Cason CL, Seidel SL, Bushmiaer M. Recovery from laparoscopic cholecystectomy procedures. AORN J. 1996 Jun;63(6):1099-103, 1106-8, 1111-2 passim. doi: 10.1016/s0001-2092(06)63296-1. PMID 8771319
- [Background] Madsen MR, Jensen KE. Postoperative pain and nausea after laparoscopic cholecystectomy. Surg Laparosc Endosc. 1992 Dec;2(4):303-5. PMID 1341550
- [Background] Dobbs FF, Kumar V, Alexander JI, Hull MG. Pain after laparoscopy related to posture and ring versus clip sterilization. Br J Obstet Gynaecol. 1987 Mar;94(3):262-6. doi: 10.1111/j.1471-0528.1987.tb02365.x. PMID 2952160
- [Background] Jackson SA, Laurence AS, Hill JC. Does post-laparoscopy pain relate to residual carbon dioxide? Anaesthesia. 1996 May;51(5):485-7. doi: 10.1111/j.1365-2044.1996.tb07798.x. PMID 8694166
- [Background] Kandil TS, El Hefnawy E. Shoulder pain following laparoscopic cholecystectomy: factors affecting the incidence and severity. J Laparoendosc Adv Surg Tech A. 2010 Oct;20(8):677-82. doi: 10.1089/lap.2010.0112. PMID 20701547
- [Background] Lee DH, Song T, Kim KH, Lee KW. Incidence, natural course, and characteristics of postlaparoscopic shoulder pain. Surg Endosc. 2018 Jan;32(1):160-165. doi: 10.1007/s00464-017-5651-5. Epub 2017 Jun 22. PMID 28643053
- [Background] Li X, Li K. Time Characteristics of Shoulder Pain after Laparoscopic Surgery. JSLS. 2021 Apr-Jun;25(2):e2021.00027. doi: 10.4293/JSLS.2021.00027. PMID 34248341
- See also: Heating pads and early mobilization for reducing postoperative shoulder pain and enhancing recovery of women undergoing gynecological laparoscopic surgery — https://fnur.stafpu.bu.edu.eg/Maternal%20and%20Newborn%20Health/1833/publications/Aziza%20Ibrahim%20Mohammed%20Hassan_B05121016_6.pdf
- See also: Ağrı kontrolünde farmakolojik olmayan yöntemler — http://dergipark.org.tr/tr/pub/hunhemsire/issue/7838/103252